CLINICAL TRIAL: NCT05072184
Title: the Effect of Erector Spinae Plane Block on Fentanyl Consumption During Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M546
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a prospective, randomized, double-blind, parallel-group clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block (Active Comparator): The patients will be randomized into two groups: ESP block group who will receive preoperative US-guided bilateral ESP block with 20 ml of bupivacaine 0.25% on each side
  Interventions: Procedure: ESP block
- Control (Sham Comparator): The patients will be randomized into two groups: ESP block group who will receive preoperative US-guided bilateral ESP block with 20 ml of saline on each side
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: ESP block — ESP block group who will receive preoperative US-guided bilateral ESP block with 20 ml of bupivacaine 0.25% on each side
  Other Names: regional anesthesia

SUMMARY:
This study aims to evaluate the effects of erector spinae plane block on intraoperative fentanyl consumption in patients undergoing abdominal hysterectomy under general anesthesia.

To our knowledge, no study in the literature demonstrates this effect.

DETAILED DESCRIPTION:
This study will be performed in Fayoum University hospital after approval of the institutional ethics committee and written informed consent. This study will be conducted as a prospective, randomized, double-blind, parallel-group clinical trial.

Inclusion criteria:

* American Society of Anesthesiologists (ASA) physical status I, II patients who will be scheduled for elective abdominal hysterectomy.
* Age range above 18.

Exclusion criteria:

* Patient refusal.
* Significant renal, hepatic and cardiovascular diseases.
* History of allergy to one of the study drugs.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders.
* Chronic opioid use, history of chronic pain and cognitive disorders.

The patients will be randomized into two groups: ESP block group who will receive preoperative US-guided bilateral ESP block with 20 ml of bupivacaine 0.25% on each side and Control group who will undergo the same procedure but with an injection of 20 ml of saline on a 1:1 ratio using a computer-generated random table. The patient's assigned group information will be elicited from a sealed opaque envelope by the anesthesiologist who will perform the ESP block and will not be involved in further data collection or patient care. The patients and both the surgical and anesthesia teams, who are responsible for patient care and data collection are blinded from the group assignments.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria:

* American Society of Anesthesiologists (ASA) physical status I, II patients who will be scheduled for elective abdominal hysterectomy.
* Age range 18-70 years

Exclusion Criteria:

* Patient refusal.

  * Significant renal, hepatic, and cardiovascular diseases.
  * History of allergy to one of the study drugs.
  * Any contraindication to regional anesthesia such as local infection or bleeding disorders.
  * Chronic opioid use, history of chronic pain and cognitive disorders.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
The total intraoperative fentanyl consumption (μg) | operative time in hours
  the total doses of intraoperative fentanyl consumption in (μg)

SECONDARY OUTCOMES:
intraoperative sevoflurane consumption (ml) | operative time in hours
  intraoperative sevoflurane consumption (ml)
post-operative fentanyl consumption in (μg) | the first 24 hours postoperative
  post-operative fentanyl consumption in the first 24 hours (μg)
VAS score | the first 24 hours postoperative
  visual analog score
mean operative times (min) | operative times in (min)
  operative times duration in (min)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
no plane

REFERENCES:
- [Background] Boules ML, Goda AS, Abdelhady MA, Abu El-Nour Abd El-Azeem SA, Hamed MA. Comparison of Analgesic Effect Between Erector Spinae Plane Block and Transversus Abdominis Plane Block After Elective Cesarean Section: A Prospective Randomized Single-Blind Controlled Study. J Pain Res. 2020 May 19;13:1073-1080. doi: 10.2147/JPR.S253343. eCollection 2020. PMID 32547172
- [Result] Azari L, Santoso JT, Osborne SE. Optimal pain management in total abdominal hysterectomy. Obstet Gynecol Surv. 2013 Mar;68(3):215-27. doi: 10.1097/OGX.0b013e31827f5119. PMID 23945838
- [Result] Hamed MA, Goda AS, Basiony MM, Fargaly OS, Abdelhady MA. Erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy: a randomized controlled study original study. J Pain Res. 2019 Apr 30;12:1393-1398. doi: 10.2147/JPR.S196501. eCollection 2019. PMID 31118757
- [Derived] Hamed MA, Boules ML, Mahmoud MAEM, Abdelghaffar RA. The effect of erector spinae plane block on fentanyl consumption during open abdominal hysterectomy: a randomised controlled study. BMC Anesthesiol. 2023 Jun 5;23(1):194. doi: 10.1186/s12871-023-02156-3. PMID 37277703